CLINICAL TRIAL: NCT01311999
Title: Surveillance and Follow-up for Latent Tuberculosis Infection and Risk of Developing Active Tuberculosis in Patients Receiving Long-term Dialysis
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201009057R
Record Dates: First submitted 2011-03-08; First posted 2011-03-10 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2013-12

CONDITIONS: To Predict the Potential of Development of Active Tuberculosis in Those Receiving Long-term Dialysis by Using Interferon-gamma Release Assy
Keywords: latent tuberculosis, renal failure, dialysis, interferon-gamma release assay
MeSH Terms: conditions — Latent Tuberculosis; Renal Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- IGRA-positive group: The subjects who have positive results of interferon-gamma release assay
- IGRA-negative group: The subjects who have negative results of interferon-gamma release assay

SUMMARY:
To follow-up the latent tuberculosis infection and the risk of developing active tuberculosis in patients receiving long-term dialysis

DETAILED DESCRIPTION:
Tuberculosis (TB) remains an important infectious disease worldwide. Taiwan is still an edemic area. In 2008, there is an incidence of 62 persons having TB per 100,000 population. To control TB, we should prevent further TB transmission via early diagnosis and treatment of latent TB. In screening the risk population for TB, patients with renal failure acquiring long-term dialysis, in addition to close contacts, have higher incidence and mortality than general population. Moreover, the risk for active TB in dialysis patients is ten to 25 times larger. In Taiwan, the dialysis group is important because it has higher prevalence (2228 per in per million people by 2009 annual report of United States Renal Data System) than other countries in the world. In particular, the dialysis patients usually has an extrapulmonary presentation for their TB, so diagnosis is always delay. Hence, we should detect latent TB in those dialysis patients for monitor them from active tuberculosis.

Currently, interferon-gamma release assays (IGRAs) are used for finding out those with latent TB and have been proven useful for those being immunocompromised, and having BCG vaccination. For dialysis patients, IGRAs have been tested and been considered better than skin tuberculin test. However, previous studied rarely observed the patients receiving peritoneal dialysis. Besides, those cross-sectional studies used the indirect evidence for diagnosis and lacked longitudinal follow-up. We thus conducted this study for observing the prevalence of latent TB in those receiving hemodialysis or peritoneal dialysis by using IGRAs. We also kept one-year follow-up for the primary outcome of active TB occurrence.

ELIGIBILITY:
Inclusion Criteria:

* age equal to or more than 18-years old
* having received dialysis more than 3 months

Exclusion Criteria:

* Positive HIV test
* Liver cirrhosis, Child-Pugh class C
* Receiving long-term systemic corticosteroid use
* Receiving chemotherapy within recent three months
* Life span is less than one year
* Being suspected to have active tuberculosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients receiving long-term dialysis
Sampling Method: Probability Sample
Enrollment: 234 (Actual)
Dates: Start 2011-02; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Development of active tuberculosis | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Chin-Chung Shu, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan